CLINICAL TRIAL: NCT00042991
Title: Phase I/II Trial of Gefitinib and Radiation in Pediatric Patients Newly Diagnosed With Brain Stem Tumors or Incompletely Resected Supratentorial Malignant Gliomas With Phase II Limited to Brain Stem Tumors
Brief Title: Gefitinib and Radiation Therapy in Treating Children With Newly Diagnosed Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03022; NCI-2012-03022 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-007 (Other: Pediatric Brain Tumor Consortium); PBTC-007 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2012-12

CONDITIONS: Untreated Childhood Anaplastic Astrocytoma; Untreated Childhood Anaplastic Oligodendroglioma; Untreated Childhood Brain Stem Glioma; Untreated Childhood Giant Cell Glioblastoma; Untreated Childhood Glioblastoma; Untreated Childhood Gliomatosis Cerebri; Untreated Childhood Gliosarcoma; Untreated Childhood Oligodendroglioma
MeSH Terms: interventions — Gefitinib; Radiotherapy; Radiation

ARMS (1):
- Treatment (gefitinib and radiation therapy) (Experimental): Phase I portion: Patients receive oral gefitinib once daily. Treatment repeats every 4 weeks for 13 courses (1 year). Patients also receive standard brain irradiation once daily, 5 days a week, for 6 weeks beginning concurrently with initiation of the first course of gefitinib. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Phase II portion: Once the MTD or the recommended Phase-II dose is determined, additional patients who have newly diagnosed BSG are treated at the MTD or the recommended Phase-II dose.
  Interventions: Drug: gefitinib; Radiation: radiation therapy; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gefitinib — Given orally
  Other Names: Iressa
Radiation: radiation therapy — Undergo standard brain irradiation
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Biological therapies such as gefitinib may interfere with the growth of the tumor cells and may make the tumor cells more sensitive to radiation therapy. This phase I/II trial is studying how well giving gefitinib together with radiation therapy works in treating children with newly diagnosed glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the safety of gefitinib administered in conjunction with irradiation in children with newly diagnosed non-disseminated diffuse intrinsic brainstem gliomas and newly diagnosed incompletely resected supratentorial malignant gliomas (STMG) not receiving enzyme inducing anticonvulsant drugs (EIACDs).

II. To define the safety of gefitinib in children with newly diagnosed, incompletely resected STMG receiving EIACDs.

III. To assess the safety and efficacy of gefitinib given with radiation therapy in children newly diagnosed with a brainstem glioma as measured by progression-free survival and to estimate the survival distribution.

SECONDARY OBJECTIVES:

I. To compare hemodynamic magnetic resonance (MR) parameters to metabolic fludeoxyglucose F 18 (FDG)-positron emission tomography (PET) scanning and correlate both with clinical response or progression in this population.

II. To characterize the expression of ErbB1 receptors in tissue from STMG patients using immunohistochemistry and western blot assays.

III. To characterize the pharmacokinetics of gefitinib in the above patient groups and determine the effects of EIACD on the pharmacokinetics.

IV. To explore the pharmacogenetic polymorphisms for gefitinib (e.g., CYP3A4/5 and BCRP) and relate them to gefitinib pharmacokinetics and pharmacodynamics (phenotype-genotype).

OUTLINE: This is a multicenter, dose-escalation study of gefitinib (Phase I closed to accrual effective 10/27/2003). Patients are stratified according to the following:

Stratum 1A: Intrinsic brain stem glioma; not receiving concurrent enzyme-inducing anticonvulsant drugs (EIACDs) Stratum 1B: Incompletely resected supratentorial malignant gliomas (STMG); not receiving concurrent EIACDs Stratum 2: Incompletely resected STMG; receiving concurrent EIACDs.

Phase I portion (patients in strata 1A, 1B, and 2) (phase I closed to accrual effective 10/27/2003): Patients receive oral gefitinib once daily. Treatment repeats every 4 weeks for 13 courses (1 year). Patients also receive standard brain irradiation once daily, 5 days a week, for 6 weeks beginning concurrently with initiation of the first course of gefitinib. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Phase II portion (patients in stratum 1A): Once the MTD or the recommended Phase-II dose is determined, additional patients who have newly diagnosed brain stem gliomas (BSG) are treated at the MTD or the recommended Phase-II dose.

Patients are followed for three months after the last protocol treatment for those enrolled strictly on the phase I component. Patients contributing to the phase II portion are followed until the earliest of date of death or three years after initiation of protocol therapy.

PROJECTED ACCRUAL: Considering the seven dose levels to be investigated in three strata, where each dose level can accrue up to six patients, a total of 126 patients (42 for each strata) may be accrued for this study within 2 years. (Phase I closed to accrual effective 10/27/2003). A total of 40 patients including the patients treated at the maximum tolerated dose or the recommended Phase-II dose during Phase I will be accrued for phase II of this study within 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Tumor:

  * Phase I: newly diagnosed non-disseminated diffuse intrinsic brainstem tumor or newly diagnosed (diagnostic scan must be within 4 weeks prior to treatment initiation), incompletely resected supratentorial malignant glioma (anaplastic astrocytoma, glioblastoma multiforme or other high-grade glioma) (STMG); the STMG group must have residual tumor evident on postoperative MRI or CT
  * Phase II: only newly diagnosed non-disseminated diffuse intrinsic brain stem glioma patients are eligible
* Performance status: Karnofsky or Lansky >= 50% assessed within two weeks prior to registration
* Prior/concurrent therapy:

  * Chemotherapy: no prior therapy allowed, including prior gefitinib treatment
  * Radiation therapy (XRT): no prior therapy allowed
  * Bone marrow transplant: none prior
  * Anti-convulsants: patients with brain stem glioma (BSG) receiving EIACD will not be eligible; patients with STMG will be eligible for this study even if they are receiving enzyme inducting anti-convulsant drugs (EIACD) and will be stratified by use of EIACDs
  * Growth factors: off all colony forming growth factor(s) > 2 weeks prior to registration (G-CSF, GM-CSF, erythropoietin)
* ANC > 1,000/ul
* Platelets > 100,000/ul (transfusion independent)
* Hemoglobin > 8g/dl (may be transfused)
* Patients may have bone marrow involvement by disease
* Creatinine < 2 x normal for age or GFR > 70 ml/min/1.73m^2
* Bilirubin < 1.5 x normal institutional normal for age
* SGPT (ALT) < 3 x institutional normal for age
* Pregnant and/or lactating patients are excluded; patients of childbearing potential should not become pregnant and should not father a child during treatment with gefitinib; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Signed informed consent according to institutional guidelines must be obtained prior to study entry

Exclusion Criteria:

* Patients with evidence of intramural hemorrhage on a scan obtained prior to enrollment or after enrollment, before treatment
* Patients with BSG must not be taking enzyme-inducing anticonvulsant drugs
* Patient must not be receiving any other anticancer or experimental drug therapy
* Patient must have no uncontrolled infection
* Patients with significant cardiac, hepatic, gastrointestinal, renal, pulmonary, or psychiatric disease are ineligible; patients with deep venous or arterial thrombosis within 6 weeks of study entry are ineligible
* Patients with disseminated disease are not permitted
* Patients with spinal disease requiring craniospinal radiation are not eligible
* Patients with completely resected supratentorial malignant gliomas patients are ineligible

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2002-07; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Geyer, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Pediatric Brain Tumor Consortium, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual to this study started with the first patient who enrolled on 07/01/2002 and ended with the last patient who enrolled on 05/31/2006. Nine institutions enrolled patients on the study.
Pre-assignment Details: There was no randomization to the three strata, which were distinct based on diagnosis and the use of enzyme inducing anti-convulsants (EIACD).
Groups:
- Stratum 1A-100 mg/m^2 of Gefitinib + Radiation: These are patients with newly diagnosed brain stem glioma who were treated at Dose 100 mg/m^2 of Gefitinib+Radiation, where Gefitinib was administered orally once daily.
- Stratum 1A-250 mg/m^2 of Gefitinib + Radiation: These are patients with newly diagnosed brain stem glioma who were treated at Dose 250 mg/m^2 of Gefitinib+Radiation, where Gefitinib was administered orally once daily.
- Stratum 1A-375 mg/m^2 of Gefitinib + Radiation: These are patients with newly diagnosed brain stem glioma who were treated at Dose 375 mg/m^2 of Gefitinib+Radiation, where Gefitinib was administered orally once daily.
- Stratum-1B: 100 mg/m^2 of Gefitinib + Radiation: These are patients with newly diagnosed, incompletely resected supertentorial malignant gliomas and NOT receiving enzyme inducing anticonvulsant drugs (EIACD), who were treated at Dose 100 mg/m^2 of Gefitinib+Radiation, where Gefitinib was administered orally once daily.
- Stratum-1B: 250 mg/m^2 of Gefitinib + Radiation: These are patients with newly diagnosed, incompletely resected supertentorial malignant gliomas and NOT receiving enzyme inducing anticonvulsant drugs (EIACD), who were treated at Dose 250 mg/m^2 of Gefitinib+Radiation, where Gefitinib was administered orally once daily.
- Stratum-1B: 375 mg/m^2 of Gefitinib + Radiation: These are patients with newly diagnosed, incompletely resected supertentorial malignant gliomas and NOT receiving enzyme inducing anticonvulsant drugs (EIACD), who were treated at Dose 375 mg/m^2 of Gefitinib+Radiation, where Gefitinib was administered orally once daily.
- Stratum-2: 100 mg/m^2 of Gefitinib + Radiation + EIACD: These are patients with newly diagnosed, incompletely resected supertentorial malignant gliomas and receiving enzyme inducing anticonvulsant drugs (EIACD), who were treated at Dose 100 mg/m^2 of Gefitinib+Radiation, where Gefitinib was administered orally once daily.
Period: Overall Study
Arm/Group | Stratum 1A-100 mg/m^2 of Gefitinib + Radiation | Stratum 1A-250 mg/m^2 of Gefitinib + Radiation | Stratum 1A-375 mg/m^2 of Gefitinib + Radiation | Stratum-1B: 100 mg/m^2 of Gefitinib + Radiation | Stratum-1B: 250 mg/m^2 of Gefitinib + Radiation | Stratum-1B: 375 mg/m^2 of Gefitinib + Radiation | Stratum-2: 100 mg/m^2 of Gefitinib + Radiation + EIACD
Started | 6 | 43 (These 43 patients form the Phase-II cohort, seven contributing from the Phase-I trial.) | 7 | 2 | 3 | 5 | 3
Phase-I Trial | 6 | 7 (These seven patients contributed to both Phase-I and Phase-II objectives.) | 7 | 2 | 3 | 5 | 3
Phase-II Trial | 0 | 36 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 1 | 0 | 0 | 0 | 1
Not Completed | 6 | 40 | 6 | 2 | 3 | 5 | 2
Not completed — Adverse Event | 1 | 4 | 2 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 2 | 0 | 1 | 0 | 0
Not completed — Disease Progression | 5 | 29 | 2 | 2 | 1 | 4 | 2
Not completed — Alternative Therapy | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1A-100 mg/m^2 of Gefitinib + Radiation | Stratum 1A-250 mg/m^2 of Gefitinib + Radiation | Stratum 1A-375 mg/m^2 of Gefitinib + Radiation | Stratum-1B: 100 mg/m^2 of Gefitinib + Radiation | Stratum-1B: 250 mg/m^2 of Gefitinib + Radiation | Stratum-1B: 375 mg/m^2 of Gefitinib + Radiation | Stratum-2: 100 mg/m^2 of Gefitinib + Radiation + EIACD | Total
Number analyzed (Participants) | 6 | 43 | 7 | 2 | 3 | 5 | 3 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 43 | 7 | 2 | 2 | 5 | 3 | 68
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.25 (2.92) | 8.02 (3.87) | 10.07 (4.71) | 9.17 (8.56) | 15.91 (5.61) | 11.69 (5.40) | 12.82 (2.37) | 9.01 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 29 | 4 | 0 | 0 | 2 | 2 | 40
  Male | 3 | 14 | 3 | 2 | 3 | 3 | 1 | 29
Region of Enrollment [Number; unit: participants]
  United States | 6 | 43 | 7 | 2 | 3 | 5 | 3 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Phase I Stratum 1A With Dose-limiting Toxicities (DLT) Observed During the First 8 Weeks of Gefitinib Therapy
Description: The dose limiting toxicity (DLT) analysis population consists of stratum 1A phase I participants who developed DLT during the maximum tolerated dose (MTD) estimation period (course 1 and 2) or who completed the MTD estimation period without DLTs. DLTs observed during courses 1 and 2 were used to estimate the MTD based on the tradional 3+3 design, where a dose is considered a safe dose only when 0 out of 3, or at most 1 out of 6 patients has DLTs. When two or more patients in a group of 2 to 6 patients had DLTs, then that dose level was considered to be too toxic.
Time Frame: Day 1 of gefitinib therapy to end of week 8
Population: This cohort includes only the patients who were enrolled and treated on Gefitinib+Radiation during the Phase I component of the trial, where the safety of Gefitinib was assedded at Dose Levels 100 mg/m^2, 250 mg/m^2, and 375 mg/m^2.
Measure: Number; unit: Participants
Groups:
- Stratum 1A-100 mg/m^2 of Gefitinib + Radiation: These are patients with brain stem glioma who were treated during the Phase-I trial of Radiation+Dose 100 mg/m^2 of Gefitinib, where Gefitinib was administered orally once daily.
- Stratum 1A-250 mg/m^2 of Gefitinib + Radiation: These are patients with brain stem glioma who were treated during the Phase-I trial of Radiation+Dose 250 mg/m^2 of Gefitinib, where Gefitinib was administered orally once daily.
- Stratum 1A-375 mg/m^2 of Gefitinib + Radiation: These are patients with brain stem glioma who were treated during the Phase-I trial of Radiation+Dose 375 mg/m^2 of Gefitinib, where Gefitinib was administered orally once daily.
Arm/Group | Stratum 1A-100 mg/m^2 of Gefitinib + Radiation | Stratum 1A-250 mg/m^2 of Gefitinib + Radiation | Stratum 1A-375 mg/m^2 of Gefitinib + Radiation
Number analyzed (Participants) | 6 | 7 | 7
Participants | 2 | 0 | 1

2. Primary Outcome: Median Progression-free Survival in Newly Diagnosed Brain Stem Gliomas
Description: Progression-free survival is defined as the interval from intiation of treatment to the earliest of disease progression (tumor increase of 25% over baseline tumor measurement; appearance of new lesion(s); or progressive/worsening neurlogical status) or death for patients who failed or to the last date of follow-up for patients without failure
Time Frame: Assessed pre-radiation, every 8 weeks for 13 courses of therapy, and then every 12 weeks
Population: Here, we only report the results for Phase-II trial as this objective was specifically for the Phase-II trial. This cohort includes seven patients who were treated during Phase-I at Dose 250 mg/m^2 of Gefitinib.
Measure: Median (Full Range); unit: Months
Groups:
- Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation: This analysis includes patients with newly diagnosed Brain Stem Glioma patients who received Dose 250 mg/m^2 of Gefitinib+Radiation.
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 43
Months | 7.43 [1.25 to 37.95]

3. Primary Outcome: Median Survival in Newly Diagnosed Brain Stem Gliomas
Description: Overall survival is defined as the interval from initiation of treatment to death or date of last contact for surviving patients
Time Frame: Assessed from the start of therapy until three years after initiation of gefitinib therapy
Measure: Median (Full Range); unit: Months
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 43
Months | 12.12 [1.71 to 37.95]

4. Secondary Outcome: Change in Tumor Volume Measured on Fluid Attenuated Inversion Recovery (FLAIR) Imaging at Before the Protocol Therapy Started and at Two Weeks After Completion of Radiation
Description: This study attempted to investigate in an exploratory manner the effect of treatment on changes in various neuroimaging variables. In this particular objective, the study aimed to investigate how radiation+gefitinib affect the tumor volume. Tumor volume is measured using Fluid Attenuated Inversion Recovery (FLAIR) before and after the radiation therapy.
Time Frame: Baseline and two weeks post completion of radiation
Population: Out of 43 patients, 35 patients had brain MRI before the treatment started and at the time of the completion of Radiation therapy. Therefore, this analysis is based on the volumetric data from these 35 patients.
Measure: Median (Full Range); unit: cc
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 35
cc | -14.03 [-48.64 to 30.56]
Statistical Analysis 1: Comparison: Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in Volume Enhancing at Two Weeks After Completion of Radiation
Description: This study attempted to investigate in an exploratory manner the effect of treatment on changes in various neuroimaging variables. Neuroimaging changes may have some association with outcome (response,survival, etc.). Volume enhancing is one parameter obtained from standard magnetic resonance imaging (MRI) studies of the brain.
Time Frame: Baseline and two weeks post completion of radiation
Population: Out of 43 patients, for only 19 patients, enhacing tumor was greater than zero based on brain MRI scans before the treatment started and at the time of the completion of Radiation therapy. Therefore, this analysis is based on the enhancing volumetric data from these 19 patients.
Measure: Median (Full Range); unit: cc
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 19
cc | 0.35 [-2.97 to 7.31]
Statistical Analysis 1: Comparison: Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation; 19 patients had Enhancing tumor at both Baseline and Post-RT time points. Thus, the following test was based on these 19 patients; Test type: Superiority or Other; p = 0.0546, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline in Diffusion Ratio at Two Weeks After Completion of Radiation
Description: This study attempted to investigate in an exploratory manner the effect of treatment on changes in various neuroimaging variables. Neuroimaging changes may have some association with outcome (response,survival, etc.). Diffusion ratio is one parameter obtained from standard magnetic resonance imaging (MRI) studies of the brain.
Time Frame: Baseline and two weeks post completion of radiation
Population: Out of 43 patients, 29 patients had diffusion scans before the treatment started and at the time of the completion of Radiation therapy. Therefore, this analysis is based on the volumetric data from these 29 patients.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 29
Ratio | -0.41 [-1.38 to 0.39]
Statistical Analysis 1: Comparison: Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change From Baseline in Perfusion Ratio at Two Weeks After Completion of Radiation
Description: This study attempted to investigate in an exploratory manner the effect of treatment on changes in various neuroimaging variables. Neuroimaging changes may have some association with outcome (response,survival, etc.). Perfusion ratio is one parameter obtained from standard magnetic resonance imaging (MRI) studies of the brain.
Time Frame: Baseline and two weeks post completion of radiation
Population: Out of 43 patients, 20 patients had perfusion scans before the treatment started and at the time of the completion of Radiation therapy. Therefore, this analysis is based on the volumetric data from these 20 patients.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 20
Ratio | 0.72 [-11.09 to 4.68]
Statistical Analysis 1: Comparison: Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Mean Tumor to Gray Matter Ratio Measured at Baseline
Description: This study attempts to characterize neuroimaging parameters from positron emission tomography. For each patient, the axial image through the tumor containing the maximum activity per pixel corresponding to the highest FluoroDeoxyGlucose (FDG) uptake was identified and a region of interest (ROI) was drawn based on the FDG definition of the tumor. The mean pixel values within the tumor ROI were normalized by those for normal gray matter to provide ratios of tumor/gray matter. Each patient has a mean tumor to gray matter ratio value and the median of these values across patients is reported.
Time Frame: Baseline
Population: Out of 43 patients, only 18 Patients had baseline PET scans. Therefore, this analysis is based on these 18 patients.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 18
Ratio | 0.55 [0.38 to 0.83]

9. Secondary Outcome: Mean Tumor to White Matter Ratio Measured at Baseline
Description: This study attempts to characterize neuroimaging parameters from positron emission tomography. For each patient, the axial image through the tumor containing the maximum activity per pixel corresponding to the highest FluoroDeoxyGlucose (FDG) uptake was identified and a region of interest (ROI) was drawn based on the FDG definition of the tumor. The mean pixel values within the tumor ROI were normalized by those for normal white matter to provide ratios of tumor/gray matter. Each patient has a mean tumor to white matter ratio value and the median of these values across patients is reported.
Time Frame: Baseline
Population: Out of 43 patients, only 18 Patients had baseline PET scans. Therefore, this analysis is based on these 18 patients.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Stratum 1A-Dose 250 mg/m^2 of Gefitinib+Radiation
Number analyzed (Participants) | 18
Ratio | 1.16 [0.92 to 2.53]

10. Secondary Outcome: Peak Serum Concentration of Gefitinib (Cmax)
Time Frame: Week 2 of course 1
Population: PK Data was combined at each dose level accross strata (Stratum 1A, Stratum 1B, and Stratum 2); at Dose 250 mg/m^2 of Gefitinib accross strata, PK data from Phase-I patients was analysed earlier for the publication of the Phase-I trial. PK data for the Phase-II patients was analyzed separately for the Phase-II publication.
Measure: Median (Full Range); unit: mcg/ml
Groups:
- Dose 250 mg/m^2 of Gefitinib (Phase II, Brain Stem Gliomas): Brain Stem Glioma patients treated on the Phase-II trial. Seven patients were treated during Phase-I at the Phase-II dose, and thus eligible for the Phase-II trial, and included in this part of the report. Only 18 patients had samples for the PK evaluation.
- Dose 250 mg/m^2 of Gefitinib (Phase I): This cohort includes all Phase-I patients treated at 250 mg/m^2 of Gefitinib regardless of diagnosis; that is, this group includes both brain stem gliomas and supratentorial malignant gliomas. Only six of 11 patients had adequate PK samples for the PK evaluation.
- Dose 100 mg/m^2 of Gefitinib: This cohort includes all Phase-I patients treated at 100 mg/m^2 of Gefitinib regardless of diagnosis; that is, this group includes both brain stem gliomas and supratentorial malignant gliomas. Eight (8) of 10 patients had adequate PK samples for the PK evaluation.
- Dose 375 mg/m^2 of Gefitinib: This cohort includes all Phase-I patients treated at 375 mg/m^2 of Gefitinib regardless of diagnosis; that is, this group includes both brain stem gliomas and supratentorial malignant gliomas. Eight of 12 patients had adequate PK samples for the PK evaluation.
Arm/Group | Dose 250 mg/m^2 of Gefitinib (Phase II, Brain Stem Gliomas) | Dose 250 mg/m^2 of Gefitinib (Phase I) | Dose 100 mg/m^2 of Gefitinib | Dose 375 mg/m^2 of Gefitinib
Number analyzed (Participants) | 18 | 6 | 8 | 8
mcg/ml | 1.10 [0.39 to 1.86] | 0.83 [0.45 to 1.36] | 0.44 [0.28 to 0.71] | 1.89 [0.93 to 2.42]

11. Secondary Outcome: Elimination Half Life of Gefitinib (t1/2)
Time Frame: Week 2 of course 1
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | Dose 250 mg/m^2 of Gefitinib (Phase II, Brain Stem Gliomas) | Dose 250 mg/m^2 of Gefitinib (Phase I) | Dose 100 mg/m^2 of Gefitinib | Dose 375 mg/m^2 of Gefitinib
Number analyzed (Participants) | 18 | 6 | 8 | 8
hour | 15.2 [9.2 to 24.9] | 17.6 [4.8 to 41.3] | 9.9 [1.8 to 19.9] | 10.4 [3.8 to 39.2]

12. Secondary Outcome: Clearance of Gefitinib (Cl)
Time Frame: Week 2 of course 1
Population: as for outcome 10
Measure: Median (Full Range); unit: L/hr/m2
Arm/Group | Dose 250 mg/m^2 of Gefitinib (Phase II, Brain Stem Gliomas) | Dose 250 mg/m^2 of Gefitinib (Phase I) | Dose 100 mg/m^2 of Gefitinib | Dose 375 mg/m^2 of Gefitinib
Number analyzed (Participants) | 18 | 6 | 8 | 8
L/hr/m2 | 15.2 [9.2 to 24.9] | 20.9 [12.6 to 33.9] | 12.8 [1.8 to 21.8] | 15.0 [5.8 to 25.8]

13. Secondary Outcome: Time of Maximum Clearance of Gefitinib (Tmax)
Time Frame: Week 2 of course 1
Population: as for outcome 10
Measure: Median (Full Range); unit: Hour
Arm/Group | Dose 250 mg/m^2 of Gefitinib (Phase II, Brain Stem Gliomas) | Dose 250 mg/m^2 of Gefitinib (Phase I) | Dose 100 mg/m^2 of Gefitinib | Dose 375 mg/m^2 of Gefitinib
Number analyzed (Participants) | 18 | 6 | 8 | 8
Hour | 3.2 [2.0 to 6.5] | 4.2 [2.0 to 6.0] | 4.9 [1.2 to 6.2] | 4.2 [2.3 to 6.4]

14. Secondary Outcome: Gefitinib Area Under the Concentration Curve From 0-24 Hours (AUC)
Time Frame: Week 2 of course 1
Population: as for outcome 10
Measure: Median (Full Range); unit: mcg/L*hr
Arm/Group | Dose 250 mg/m^2 of Gefitinib (Phase II, Brain Stem Gliomas) | Dose 250 mg/m^2 of Gefitinib (Phase I) | Dose 100 mg/m^2 of Gefitinib | Dose 375 mg/m^2 of Gefitinib
Number analyzed (Participants) | 18 | 6 | 8 | 8
mcg/L*hr | 16.4 [10.0 to 27.1] | 11.8 [4.3 to 16.7] | 5.3 [3.7 to 11.8] | 25.3 [18.4 to 35.3]

15. Secondary Outcome: Number of Patients With Epidermal Growth Factor Receptor (EGFR) Amplification
Description: Epidermal growth factor receptor (EFGR) is a protein found on the surface of cells to which epidermal growth factor (EGF) binds. When EGF attaches to EGFR, it activates the enzyme tyrosine kinase, triggering reactions that cause the cells to grow and multiply.
Time Frame: Pre-treatment
Population: Epidermal growth factor receptor is only possible with tumor sample, which is only potentially available from supratentorial malignant glioma patients treated on Stratum-1B and Stratum-2. Of 10 Stratum-1B and 3 Stratum-2 patients (n=13), tumor material was available from 11 patients (8 in Stratum-1A and 3 in Stratum-2).
Measure: Number; unit: Participants
Groups:
- Stratum IB and Stratum II: Activation and mutations of EGFR have been associated with many cancers. In this secondary objective, we identify how many patients have activated EGFR and this requires a tumor sample from patients, which is only available from supratentorial malignant glioma patients treated on Stratum IB and Stratum II.
Arm/Group | Stratum IB and Stratum II
Number analyzed (Participants) | 11
Participants | 5

ADVERSE EVENTS:
Groups:
- Stratum IA at Dose 100 mg/m^2: Brain Stem Glioma patients treated at 100 mg/m2
- Stratum IA at Dose 250 mg/m^2: Brain Stem Glioma patients treated at 250 mg/m2
- Stratum IA at Dose 375 mg/m^2: Brain Stem Glioma patients treated at 375 mg/m2
- Stratum IB at Dose 100 mg/m^2: Patients with STMG treated at 100 mg/m2
- Stratum IB at Dose 250 mg/m^2: Patients with STMG treated at 250 mg/m2
- Stratum IB at Dose 375 mg/m^2: Patients with STMG treated at 375 mg/m2
- Stratum II at Dose 100 mg/m^2: Patients with STMG treated at 100 mg/m2 who are receiving EIACD
Arm/Group | Stratum IA at Dose 100 mg/m^2 | Stratum IA at Dose 250 mg/m^2 | Stratum IA at Dose 375 mg/m^2 | Stratum IB at Dose 100 mg/m^2 | Stratum IB at Dose 250 mg/m^2 | Stratum IB at Dose 375 mg/m^2 | Stratum II at Dose 100 mg/m^2
Serious Adverse Events (participants affected / at risk) | 2/6 | 15/43 | 5/7 | 1/2 | 1/3 | 5/5 | 1/3
Other Adverse Events (participants affected / at risk) | 6/6 | 43/43 | 7/7 | 2/2 | 3/3 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum IA at Dose 100 mg/m^2 (N=6) | Stratum IA at Dose 250 mg/m^2 (N=43) | Stratum IA at Dose 375 mg/m^2 (N=7) | Stratum IB at Dose 100 mg/m^2 (N=2) | Stratum IB at Dose 250 mg/m^2 (N=3) | Stratum IB at Dose 375 mg/m^2 (N=5) | Stratum II at Dose 100 mg/m^2 (N=3)
Anorexia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Bilirubin (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CNS hemorrhage/bleeding (Nervous system disorders) | 0 | 3 | 1 | 0 | 1 | 2 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Death not associated with CTCAE term (Disease progression NOS ) (General disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Dehydration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diarrhea patients without colostomy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (lethargy, malaise, asthenia) (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 3 | 0
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils (Bladder (urinary) ) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils (Conjunctiva ) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils (Skin (cellulitis) ) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection with unknown ANC (Brain (encephalitis, infectious) ) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection without neutropenia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 0 | 1 | 2 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurology - Other (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy - cranial (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neuropathy - sensory (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neuropathy: cranial (CN IX Motor-pharynx; Sensory-ear, pharynx, tongue ) (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Speech impairment (e.g., dysphasis or aphasia) (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Weight loss (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibrinogen (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum IA at Dose 100 mg/m^2 (N=6) | Stratum IA at Dose 250 mg/m^2 (N=43) | Stratum IA at Dose 375 mg/m^2 (N=7) | Stratum IB at Dose 100 mg/m^2 (N=2) | Stratum IB at Dose 250 mg/m^2 (N=3) | Stratum IB at Dose 375 mg/m^2 (N=5) | Stratum II at Dose 100 mg/m^2 (N=3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 | 22 | 2 | 0 | 1 | 1 | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 | 13 | 1 | 0 | 1 | 1 | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 | 15 | 2 | 1 | 1 | 3 | 0
Alkaline phosphatase (Investigations) | 0 | 4 | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 1 | 0 | 0 | 2 | 0
Amylase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 11 | 1 | 1 | 1 | 0 | 1
Ataxia (incoordination) (Nervous system disorders) | 3 | 10 | 2 | 1 | 0 | 0 | 1
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 | 5 | 2 | 0 | 0 | 0 | 0
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 | 20 | 3 | 0 | 2 | 2 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 18 | 2 | 0 | 1 | 1 | 0
Constitutional Symptoms - Other (Specify, __) (General disorders) | 5 | 4 | 7 | 2 | 3 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 14 | 0 | 0 | 0 | 2 | 0
Creatinine (Investigations) | 0 | 3 | 1 | 0 | 0 | 0 | 0
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 4 | 14 | 1 | 0 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 0 | 5 | 1 | 0 | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 26 | 2 | 0 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0
Dry eye syndrome (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 17 | 3 | 0 | 0 | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 22 | 0 | 0 | 0 | 0 | 0
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 | 13 | 1 | 0 | 0 | 1 | 0
Fibrinogen (Investigations) | 1 | 3 | 2 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 | 16 | 4 | 1 | 1 | 4 | 1
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4 | 8 | 2 | 0 | 0 | 1 | 0
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 | 15 | 0 | 0 | 1 | 2 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 | 4 | 1 | 0 | 0 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 4 | 12 | 4 | 0 | 0 | 1 | 1
Hot flashes/flushes (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incontinence, urinary (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Infection - Other (Specify, __) (Infections and infestations) | 5 | 7 | 2 | 0 | 3 | 3 | 1
Insomnia (Psychiatric disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytes (total WBC) (Investigations) | 4 | 19 | 3 | 2 | 1 | 2 | 1
Lymphopenia (Investigations) | 5 | 25 | 4 | 0 | 1 | 3 | 0
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 | 10 | 1 | 0 | 1 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Metabolic/Laboratory - Other (Specify, __) (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 17 | 3 | 1 | 1 | 3 | 0
Neurology - Other (Specify, __) (Nervous system disorders) | 1 | 5 | 2 | 0 | 1 | 2 | 1
Neuropathy: motor (Nervous system disorders) | 3 | 12 | 4 | 0 | 1 | 0 | 1
Neuropathy: sensory (Nervous system disorders) | 2 | 3 | 0 | 1 | 0 | 2 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 | 8 | 2 | 1 | 1 | 1 | 1
Nystagmus (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ocular surface disease (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 | 3 | 0 | 1 | 1 | 0 | 0
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 21 | 4 | 1 | 1 | 0 | 1
Platelets (Investigations) | 2 | 6 | 1 | 0 | 0 | 2 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 6 | 1 | 1 | 0 | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 20 | 2 | 1 | 0 | 2 | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 | 29 | 5 | 0 | 2 | 2 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 7 | 0 | 0 | 0 | 0 | 0
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 2 | 5 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 | 10 | 4 | 0 | 1 | 1 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 10 | 4 | 0 | 1 | 1 | 0
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 | 6 | 0 | 0 | 0 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 32 | 4 | 2 | 2 | 3 | 0
Weight gain (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less